CLINICAL TRIAL: NCT01868230
Title: Proyecto Mama: Lifestyle Intervention in Overweight and Obese Pregnant Hispanic Women
Brief Title: Lifestyle Intervention in Overweight and Obese Pregnant Hispanic Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of California, San Diego (Other); Northeastern University (Other); Baystate Medical Center (Other)
Responsible Party: Principal Investigator, Lisa Chasan-Taber, Professor of Epidemiology, University of Massachusetts, Amherst
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01DK097011-01A1 (NIH); 1R01DK097011-01A1 (NIH)
Record Dates: First submitted 2013-05-29; First posted 2013-06-04 (Estimated); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle Intervention (Experimental): Stage-matched physical activity and diet intervention materials and health education.
  Interventions: Behavioral: Lifestyle Intervention
- Health and Wellness (No Intervention): HW served as the comparison group and received the same number of in-person sessions, telephone calls, and mailings at the same time points as LI. Content was limited to general information available to the public from the ACOG and the American Academy of Pediatrics and did not mention exercise behavior change.

INTERVENTIONS:
Behavioral: Lifestyle Intervention
  Arms: Lifestyle Intervention

SUMMARY:
The overall goal of this randomized controlled trial is to test the efficacy of a culturally and linguistically modified, individually tailored lifestyle intervention to reduce excess gestational weight gain (GWG), increase postpartum weight loss, and improve maternal metabolic status among overweight/obese Hispanic women.

DETAILED DESCRIPTION:
The overall goal of this randomized controlled trial is to test the efficacy of a culturally and linguistically modified, individually tailored lifestyle intervention to reduce excess gestational weight gain (GWG), increase postpartum weight loss, and improve maternal metabolic status among overweight/obese Hispanic women. Specific aims are to evaluate the impact of the intervention on 1) GWG and postpartum weight loss, 2) pregnancy and postpartum biomarkers of insulin resistance (i.e., glucose, insulin, HbA1c, HOMA, leptin, adiponectin), 3) postpartum biomarkers of cardiovascular risk (i.e., blood lipids, blood pressure), 4) offspring outcomes (i.e., anthropometric measures and biomarkers of insulin resistance), and 5) to evaluate the cost-effectiveness of the intervention per average incremental improvement in the outcome variables. Overweight/obese Hispanic women will be recruited in early pregnancy (around 10 wks gestation) and randomly assigned to a Lifestyle Intervention (n=150) or a Comparison Health and Wellness (control) Intervention (n=150). The intervention will utilize exercise (R01NR011295) and dietary intervention materials (R18DK067549) culturally adapted for Hispanics and shown to be efficacious in our previous controlled trials in this ethnic group. Multimodal contacts (i.e., in-person, telephone counseling, and mailed print-based materials) will be used to deliver the intervention during pregnancy (~12 wks gestation to delivery) continuing into postpartum (~6 wks to 6 mos postpartum); follow-up will continue for one year postpartum. Targets of the intervention are to achieve Institute of Medicine Guidelines for GWG and postpartum weight loss; ACOG guidelines for physical activity through increasing walking and developing a more active lifestyle; and reduction in total calories by following a balanced healthy diet in compliance with American Diabetes Association guidelines. The intervention draws from Social Cognitive Theory and the Transtheoretical Model and includes strategies for partner and/or family support to address the specific social, cultural, and economic challenges faced by underserved Hispanic women. Measures of compliance will include actigraphs and Hispanic food frequency questionnaires. The proposed project builds upon the expertise of the investigative team in conducting randomized controlled trials of exercise interventions among Hispanic pregnant women (R01 DK074876) and dietary interventions among low-income Hispanics with type 2 diabetes (R18 DK0658850) and can readily be translated into clinical practice in underserved and minority populations.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic women
* Overweight or obese before pregnancy (BMI >25 kg/m2)
* 16-45 years old

Exclusion Criteria:

* prepregnancy BMI <25 kg/m2
* history of type 2 diabetes, heart disease, or chronic renal disease
* contraindications to postpartum participation in moderate physical activity or a low-fat/high-fiber diet (e.g., Crohn's disease, ulcerative colitis)
* inability to read English or Spanish at a 6th grade level
* >16 wks gestation
* current medications which adversely influence glucose tolerance
* not planning to continue to term or deliver at the study site
* pregnant with twins or triplets

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 232 (Actual)
Dates: Start 2014-06; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Chasan-Taber, ScD, Principal Investigator — University of Massachusetts, Amherst
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gubrium A, Leckenby D, Harvey MW, Marcus BH, Rosal MC, Chasan-Taber L. Perspectives of health educators and interviewers in a randomized controlled trial of a postpartum diabetes prevention program for Latinas: a qualitative assessment. BMC Health Serv Res. 2019 Jun 6;19(1):357. doi: 10.1186/s12913-019-4207-x. PMID 31170973
- [Derived] Chasan-Taber L, Marcus BH, Rosal MC, Tucker KL, Hartman SJ, Pekow P, Stanek E 3rd, Braun B, Solomon CG, Manson JE, Goff SL, Markenson G. Proyecto Mama: a lifestyle intervention in overweight and obese Hispanic women: a randomised controlled trial--study protocol. BMC Pregnancy Childbirth. 2015 Jul 30;15:157. doi: 10.1186/s12884-015-0575-3. PMID 26223246

RESULTS

PARTICIPANT FLOW:
Groups:
- Lifestyle Intervention: Stage-matched physical activity and diet intervention materials and health education.
  Lifestyle Intervention
Period: Overall Study
Arm/Group | Lifestyle Intervention | Health and Wellness
Started | 74 | 74
6 Week Postpartum Data | 35 | 41
6 Month Postpartum Data | 20 | 33
12 Months Postpartum | 22 | 24
Completed | 74 | 74
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The primary analysis involved an intent-to-treat analysis among all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Intervention | Health and Wellness | Total
Number analyzed (Participants) | 74 | 74 | 148
Age, Categorical [Count of Participants; unit: Participants] — Population: The primary analysis involved an intent-to-treat analysis among all randomized participants.
  Participants
    <=18 years | 10 | 11 | 21
    Between 18 and 65 years | 64 | 63 | 127
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The primary analysis involved an intent-to-treat analysis among all randomized participants.
  Participants
    Female | 74 | 74 | 148
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The primary analysis involved an intent-to-treat analysis among all randomized participants.
  Participants
    Hispanic or Latino | 74 | 74 | 148
    Not Hispanic or Latino | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: The primary analysis involved an intent-to-treat analysis among all randomized participants.
  participants
    United States | 74 | 74 | 148
BMI [Mean (Standard Deviation); unit: kg/m2] — Population: The primary analysis involved an intent-to-treat analysis among all randomized participants.
  kg/m2 | 33.8 (6.7) | 33.3 (7.6) | 33.5 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Gestational Weight Gain
Description: Gestational weight change will be measured as the difference between weight at delivery and prepregnancy weight as abstracted from the medical record. The analysis involved an intent-to-treat analysis among the entire sample of randomized participants. Missing postpartum weights were imputed in the manner of prior weight loss trials with the use of 10 random multivariate imputations based on observed variables at baseline.
Time Frame: delivery
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 74 | 74
kg | 7.9 [4.9 to 11.0] | 10.4 [7.4 to 13.3]

2. Primary Outcome: Postpartum Weight Change
Description: Postpartum weight change will be measured as the difference between weight at 6 or 12 mos postpartum and weight at delivery. Weight will be measured on a digital scale. The analysis involved an intent-to-treat analysis among the entire sample of randomized participants. Missing postpartum weights were imputed in the manner of prior weight loss trials with the use of 10 random multivariate imputations based on observed variables at baseline.
Time Frame: 6 weeks postpartum, 6 months postpartum, 12 months postpartum
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 74 | 74
kg
  6 weeks postpartum | 3.2 [0.2 to 6.2] | 3.2 [0.8 to 5.6]
  6 months postpartum | 3.9 [0.3 to 7.5] | 5.7 [2.2 to 9.1]
  12 months postpartum | 6.4 [1.0 to 11.9] | 8.4 [3.6 to 13.2]

3. Primary Outcome: Percent of Participants Meeting Postpartum Weight Goals
Description: Postpartum weight goals will be defined as a 5% reduction from prepregnancy weight. Weight will be measured on a digital scale. The analysis involved an intent-to-treat analysis among the entire sample of randomized participants. Missing postpartum weights were imputed in the manner of prior weight loss trials with the use of 10 random multivariate imputations based on observed variables at baseline.
Time Frame: 6 weeks postpartum, 6 months postpartum, 12 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 74 | 74
Participants
  6 weeks postpartum | 12 | 9
  6 months postpartum | 12 | 7
  12 months postpartum | 12 | 6

4. Primary Outcome: Fasting Glucose (FG)
Description: Fasting Glucose (FG) will be measured enzymatically on the Roche P Modular system using Roche Diagnostics reagents (Indianapolis, IN)(mg/dL). The analysis involved an intent-to-treat analysis among the entire sample of randomized participants.
Time Frame: 6 weeks postpartum, 6 months postpartum, 12 months postpartum
Population: Biomarker data not provided by the remainder of participants.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 51 | 58
mg/dL
  6 wks postpartum | 85.22 (9.77) | 83.89 (11.39)
  6 mos postpartum | 87.41 (13.71) | 84.92 (14.64)
  12 mos postpartum | 87.41 (8.16) | 91.52 (12.47)

5. Primary Outcome: Fasting Insulin
Description: Fasting Insulin (FI) will be measured by an electrochemiluminescence immunoassay on the Roche E Modular system in uU/mL. The analysis involved an intent-to-treat analysis among the entire sample of randomized participants.
Time Frame: 6 weeks postpartum, 6 months postpartum, 12 months postpartum
Population: Biomarker data not provided by the remainder of participants.
Measure: Mean (Standard Deviation); unit: iU/mL
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 51 | 58
iU/mL
  6 wks postpartum | 14.65 (7.65) | 20.57 (21.40)
  6 mos postpartum | 21.37 (18.38) | 26.53 (16.22)
  12 mos postpartum | 16.67 (8.83) | 21.54 (16.86)

6. Primary Outcome: Hemoglobin A1c (HbA1c)
Description: The Hemoglobin A1c (HbA1c) determination on the Roche P Modular system will be based on turbidimetric immunoinhibition using packed red cells. The analysis involved an intent-to-treat analysis among the entire sample of randomized participants.
Time Frame: 6 weeks postpartum, 6 months postpartum, 12 months postpartum
Population: Biomarker data not provided by the remainder of participants.
Measure: Mean (Standard Deviation); unit: % of HbA1c
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 51 | 58
% of HbA1c
  6 wks postpartum | 5.08 (0.29) | 5.04 (0.35)
  6 mos postpartum | 5.19 (0.31) | 5.20 (0.26)
  12 mos postpartum | 5.18 (0.33) | 5.13 (0.31)

7. Primary Outcome: Adiponectin
Description: Total Adiponectin (Multimeric) will be measured using an ELISA method from ALPCO Diagnostics Inc. (Salem, NH). The analysis involved an intent-to-treat analysis among the entire sample of randomized participants.
Time Frame: 6 weeks postpartum, 6 months postpartum, 12 months postpartum
Population: Biomarker data not provided by the remainder of participants.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 51 | 58
ng/ml
  6 wks postpartum | 3.19 (1.63) | 3.41 (1.71)
  6 mos postpartum | 3.18 (1.64) | 2.94 (1.76)
  12 mos postpartum | 3.09 (1.54) | 3.55 (2.07)

8. Primary Outcome: Total Leptin
Description: Leptin will be measured by an ultra-sensitive ELISA assay, an enzymatically amplified "two-step" sandwich-type immunoassay (R&D Systems, Minneapolis, MN) (pg/mL). The analysis involved an intent-to-treat analysis among the entire sample of randomized participants.
Time Frame: 6 weeks postpartum, 6 months postpartum, 12 months postpartum
Population: Biomarker data not provided by the remainder of participants.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 51 | 58
pg/mL
  6 wks postpartum | 44.51 (16.34) | 50.13 (22.24)
  6 mos postpartum | 44.64 (28.97) | 52.28 (29.99)
  12 mos postpartum | 42.44 (21.37) | 42.39 (16.19)

9. Primary Outcome: Total Cholesterol
Description: Lipoprotein Profile: will be simultaneously performed on the Roche P Modular system. Total Cholesterol will be measured enzymatically (mg/dL). The analysis involved an intent-to-treat analysis among the entire sample of randomized participants.
Time Frame: 6 weeks postpartum, 6 months postpartum, 12 months postpartum
Population: Biomarker data not provided by the remainder of the randomized participants.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 51 | 58
mg/dL
  6 wks postpartum | 167.75 (28.61) | 162.28 (34.79)
  6 mos postpartum | 165.18 (26.52) | 153.96 (27.81)
  12 mos postpartum | 164.41 (23.00) | 147.29 (24.83)

10. Primary Outcome: Low Density Lipoprotein Cholesterol
Description: Low Density Lipoprotein Cholesterol will be determined by a homogenous direct method (mg/dL).The analysis involved an intent-to-treat analysis among the entire sample of randomized participants.
Time Frame: 6 weeks postpartum, 6 months postpartum, 12 months postpartum
Population: Biomarker data not provided by the remainder of the randomized participants.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 51 | 58
mg/dL
  6 wks postpartum | 108.27 (29.57) | 101.03 (29.00)
  6 mos postpartum | 103.85 (23.21) | 96.52 (26.49)
  12 mos postpartum | 105.79 (24.35) | 91.60 (22.76)

11. Primary Outcome: High Density Lipoprotein Cholesterol.
Description: The concentration of High Density Lipoprotein Cholesterol will be determined using a direct enzymatic colorimetric assay (mg/dL). The analysis involved an intent-to-treat analysis among the entire sample of randomized participants.
Time Frame: 6 weeks postpartum, 6 months postpartum, 12 months postpartum
Population: Biomarker data not provided by the remainder of the randomized participants.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 51 | 58
mg/dL
  6 wks postpartum | 42.75 (6.85) | 43.50 (9.45)
  6 mos postpartum | 48.12 (19.91) | 42.04 (8.58)
  12 mos postpartum | 47.53 (11.54) | 42.52 (10.72)

12. Primary Outcome: Triglycerides
Description: Triglycerides will be measured enzymatically with correction for endogenous glycerol (mg/dL). The analysis involved an intent-to-treat analysis among the entire sample of randomized participants.
Time Frame: 6 weeks postpartum, 6 months postpartum, 12 months postpartum
Population: Biomarker data not provided by the remainder of the randomized participants.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 51 | 58
mg/dL
  6 wks postpartum | 94.08 (49.30) | 101.94 (49.34)
  6 mos postpartum | 99.19 (61.02) | 92.73 (45.86)
  12 mos postpartum | 88.38 (35.98) | 85.90 (46.17)

13. Primary Outcome: High Sensitivity C-Reactive Protein
Description: The concentration of High Sensitivity C-Reactive Protein (hsCRP) will be determined using an immunoturbidimetric assay on the Roche P Modular system using reagents and calibrators from DiaSorin (Stillwater, MN) (mg/L). The analysis involved an intent-to-treat analysis among the entire sample of randomized participants.
Time Frame: 6 weeks postpartum, 6 months postpartum, 12 months postpartum
Population: Biomarker data not provided by the remainder of the randomized participants.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 51 | 58
mg/L
  6 wks postpartum | 4.63 (3.98) | 7.02 (10.63)
  6 mos postpartum | 6.62 (9.39) | 7.08 (8.50)
  12 mos postpartum | 6.48 (6.85) | 5.50 (5.65)

14. Primary Outcome: Compliance With IOM Weight Gain Guidelines for Pregnancy.
Description: Compliance with IOM weight gain guidelines during pregnancy is measured by comparing the observed gestational weight gain (GWG) with the 2009 IOM Guidelines. The analysis involved an intent-to-treat analysis among the entire sample of randomized participants. Missing weights were imputed in the manner of prior trials with the use of 10 random multivariate imputations based on observed variables at baseline. Total GWG was calculated by subtracting pre-pregnancy weight from weight at delivery and was categorized as "below," "within," or "above" IOM guidelines based on the IOM's 2009 GWG guidelines: specifically, women with an underweight BMI are advised to gain a total of 28-40 lbs, women with a BMI in the normal weight category are advised to gain 25-35 lbs., women with a BMI in the overweight category are advised to gain 15-25 lbs, and women with a BMI in the obese category are advised to gain 11-20 lbs.
Time Frame: delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 74 | 74
Participants
  Below IOM Guidelines | 13 | 12
  Within IOM Guidelines | 9 | 13
  Above IOM Guidelines | 41 | 45
  missing | 11 | 4

15. Primary Outcome: Child Waist Circumference
Description: measuring tape
Time Frame: delivery
Population: Anthropometric measures not available for the remainder of the randomized participants.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 21 | 21
cm | 41 (4.5) | 41 (4.49)

16. Primary Outcome: Child Head Circumference
Description: measuring tape
Time Frame: delivery
Population: Anthropometric measures not available for the remainder of the randomized participants.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 19 | 19
cm | 55 (4.6) | 54.9 (4.5)

17. Primary Outcome: Child Skinfold Thicknesses - Subcapsular and Triceps
Description: calipers
Time Frame: delivery
Population: Anthropometric measures not available for the remainder of the randomized participants.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 19 | 19
mm
  subcapsular | 8.8 (2.5) | 9.1 (2.4)
  triceps | 10.4 (10.1) | 10.1 (2.9)

18. Primary Outcome: Fetal Growth
Description: Birthweight-for-gestational age z-scores will be calculated by subtracting the mean and dividing by the standard deviation from a standardization population (specifically, the 2014 Natality data from National Center for Health Statistics using data limited to Hispanic ethnicity). A Z-score of 0 represents the population mean. Z score values <0 represent scores lower than the population average observed in the standardization population. It remains to be established which z score range (percentile and SD) is associated with optimal short- and long-term offspring health.
Time Frame: delivery
Population: Anthropometric measures not available for the remainder of the randomized participants.
Measure: Geometric Mean (Standard Deviation); unit: z score
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 21 | 21
z score | 0.21 (1.2) | -0.08 (1.2)

19. Primary Outcome: Ponderal Index
Description: The ponderal index is calculated as birth weight (g) x 100/birth length (cm). A lower ponderal index is typically used to identify neonates that were affected by intrauterine growth restriction. For example, ponderal indexes between 2.5 and 3.0 are generally considered normal, between 2.0 and 2.5 marginal, and less than 2.0 low (unhealthy).
Time Frame: delivery
Population: Anthropometric measures not available for the remainder of the randomized participants.
Measure: Mean (Standard Deviation); unit: g/m^3
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 21 | 21
g/m^3 | 3.15 (1.1) | 2.89 (0.96)

20. Primary Outcome: Birthweight
Description: scale
Time Frame: delivery
Population: Anthropometric measures not available for the remainder of the randomized participants.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 21 | 21
grams | 3300.2 (556.7) | 3247.3 (600.3)

21. Primary Outcome: Child Length
Description: measuring tape
Time Frame: delivery
Population: Anthropometric measures not available for the remainder of the randomized participants.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 21 | 22
cm | 23.5 (2.6) | 24.0 (4.2)

22. Post Hoc Outcome: Physical Activity
Description: Total activity according to intensity will be measured via the Pregnancy Physical Activity Questionnaire (PPAQ). The American College of Gynecologists (ACOG) recommend that pregnant women obtain at least 30 minutes of moderate-intensity PA on most days of the week during pregnancy and postpartum. Therefore, meeting ACOG guidelines will be defined as women who obtain at least 150 minutes of moderate to vigorous intensity activity during exercise.
Time Frame: 6 weeks postpartum, 6 months postpartum, 12 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 74 | 74
Participants
  Met ACOG PA guidelines | 24 | 31
  Did not meet ACOG PA guidelines | 50 | 43

23. Post Hoc Outcome: Alternate Healthy Eating Index-Pregnancy (AHEI-P)
Description: Total calories, along with the other nutrients, will be measured via three 24-hr dietary recalls. Alternate Healthy Eating Index-Pregnancy (AHEI-P) scores were calculated. The AHEI-P is a dietary quality index based on a 130-point scale with 0-10 points awarded for optimal intake of six food groups (vegetables; whole fruit; whole grains; sugar-sweetened beverages; nuts and legumes; red/processed meats) and seven nutrient-based categories (trans fats; long-chain fats; PUFA; Na; Ca; folate; Fe). The AHEI range is from 0 to 130 with a higher score indicative of a higher quality diet.
Time Frame: mid pregnancy (mean 14.2 [SD 4.3]) weeks gestation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Intervention | Health and Wellness
Number analyzed (Participants) | 74 | 74
units on a scale | 57.6 (13.6) | 55.6 (13.6)

ADVERSE EVENTS:
Time Frame: AE data collected at follow up visits (delivery, 6 weeks, 6 and 12 months post partum)
Arm/Group | Lifestyle Intervention | Health and Wellness
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/74
Other Adverse Events (participants affected / at risk) | 0/74 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-09): https://cdn.clinicaltrials.gov/large-docs/30/NCT01868230/Prot_SAP_000.pdf